CLINICAL TRIAL: NCT02752802
Title: Single Site Randomized Control Trial Evaluating the DyeVert System
Brief Title: DyeVert System RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TP-6495
Record Dates: First submitted 2016-04-22; First posted 2016-04-27 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Coronary Angiography
Keywords: Contrast Media; Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): The treatment group will include standard of care for diagnostic angiogram along with the utilizization of the DyeVert system.
  Interventions: Device: Diagnostic Coronary Angiogram
- Control (Active Comparator): The control group will include standard of care for diagnostic coronary angiograms.
  Interventions: Device: Diagnostic Coronary Angiogram

INTERVENTIONS:
Device: Diagnostic Coronary Angiogram — Diagnostic angiographic procedure with the use of the DyeVert System.

SUMMARY:
The purpose of this study is to evaluate the amount of contrast media (CM) saved using the DyeVert system in diagnostic angiographic procedures compared to a control group.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel group, single center clinical evaluation of the DyeVert System. Subjects undergoing a diagnostic coronary angiogram procedure with a 5 French catheter are eligible to participate in this study. The treatment group will use the DyeVert System.

The trial will be conducted at one center, located in Germany. A sample size of 96 evaluable subjects will provide a sufficient number of samples to evaluate the primary objectives.

Randomization will occur following confirmation that the subject meets the inclusion/exclusion criteria and has signed an informed consent. Subjects that are anticipated to be a diagnostic only procedure, but end up being an ad-hoc PCI, can still remain enrolled in the trial. If a subject proceeds to a PCI, data will only be collected through the diagnostic portion of the case.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is indicated for a diagnostic coronary angiogram procedure with a 5 French catheter only.
2. The subject is ≥ 18 years of age
3. The subject is willing and able to provide appropriate informed consent.

Exclusion Criteria:

1. Subject is undergoing a STEMI procedure
2. Subject has previously been diagnosed with anomalous coronary anatomy
3. Subject has previously underwent coronary artery bypass grafting
4. Subject has severe peripheral artery disease at access site
5. Subject is having a staged PCI
6. The subject is female and currently pregnant
7. In the investigator's opinion, the subject is not considered to be a suitable candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Desch, MD, Principal Investigator — University Hospital of Schleswig-Holstein, Lubeck
Locations (1):
- University Hospital of Schleswig-Holstein, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown JR, Solomon RJ, Sarnak MJ, McCullough PA, Splaine ME, Davies L, Ross CS, Dauerman HL, Stender JL, Conley SM, Robb JF, Chaisson K, Boss R, Lambert P, Goldberg DJ, Lucier D, Fedele FA, Kellett MA, Horton S, Phillips WJ, Downs C, Wiseman A, MacKenzie TA, Malenka DJ; Northern New England Cardiovascular Disease Study Group. Reducing contrast-induced acute kidney injury using a regional multicenter quality improvement intervention. Circ Cardiovasc Qual Outcomes. 2014 Sep;7(5):693-700. doi: 10.1161/CIRCOUTCOMES.114.000903. Epub 2014 Jul 29. PMID 25074372
- [Background] Gruberg L, Mintz GS, Mehran R, Gangas G, Lansky AJ, Kent KM, Pichard AD, Satler LF, Leon MB. The prognostic implications of further renal function deterioration within 48 h of interventional coronary procedures in patients with pre-existent chronic renal insufficiency. J Am Coll Cardiol. 2000 Nov 1;36(5):1542-8. doi: 10.1016/s0735-1097(00)00917-7. PMID 11079656
- [Background] Klein LW, Sheldon MW, Brinker J, Mixon TA, Skelding K, Strunk AO, Tommaso CL, Weiner B, Bailey SR, Uretsky B, Kern M, Laskey W; Interventional Committee of the Society for Cardiovascular Angiography and Interventions. The use of radiographic contrast media during PCI: a focused review: a position statement of the Society of Cardiovascular Angiography and Interventions. Catheter Cardiovasc Interv. 2009 Nov 1;74(5):728-46. doi: 10.1002/ccd.22113. No abstract available. PMID 19830793
- [Background] Lameire N, Kellum JA; KDIGO AKI Guideline Work Group. Contrast-induced acute kidney injury and renal support for acute kidney injury: a KDIGO summary (Part 2). Crit Care. 2013 Feb 4;17(1):205. doi: 10.1186/cc11455. PMID 23394215
- [Background] Levy EM, Viscoli CM, Horwitz RI. The effect of acute renal failure on mortality. A cohort analysis. JAMA. 1996 May 15;275(19):1489-94. PMID 8622223

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 48 | 48
Completed | 47 | 48
Not Completed | 1 | 0
Not completed — Contrast Volume Not Collected | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (13.6) | 66.2 (12.8) | 67.4 (13.2)
Gender [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Total Volume of CM Used Comparing the DyeVert Group to the Control Group.
Description: DyeVert is intended to reduce the total amount of contrast media (CM) administered during procedures requiring the injection of contrast media. Clinical evidence has demonstrated that CM can be toxic to the kidneys, leading to contrast induced nephropathy (CIN)
Time Frame: All data will be collected on the day of the procedure, over an average of 12 hours.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treatment | Control
Number analyzed (Participants) | 47 | 48
ml | 38.0 (13.1) | 62.5 (12.7)

2. Secondary Outcome: Assessment of the Quality of Angiographic Images Between Groups
Description: To assess the adequacy of the image quality. The proportion of images in which contrast opacification is deemed sufficient to evaluate the desired anatomical structures adequately will be compared between the DyeVert and control groups.
Time Frame: AlAll data will be collected on the day of the procedure, over an average of 12 hours.
Measure: Count of Units; unit: Images
Units Other Than Participants: Images
Arm/Group | Control | Treatment
Number analyzed (Participants) | 48 | 48
Number analyzed (Images) | 399 | 404
Images | 379 | 386

3. Secondary Outcome: Assessment of Incidence of Serious Adverse Device Effect for Subjects Treated With the DyeVert System During the Procedure.
Description: To assess the incidence of Serious Adverse Device Effect for subjects treated with the DyeVert System during the procedure for treatment subjects only.
Time Frame: All data will be collected on the day of the procedure, over an average of 12 hours.
Population: Only treatments subjects were analyzed for this endpoint.
Measure: Number; unit: Number of Events
Arm/Group | Treatment
Number analyzed (Participants) | 48
Number of Events | 0

ADVERSE EVENTS:
Time Frame: At point of discharge from index procedure, approximetly 12 hours.
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 2/48 | 4/48
Other Adverse Events (participants affected / at risk) | 2/48 | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=48) | Control (N=48)
Extended Hospital Stay (General disorders) | 2 (2) | 2 (2)
Death (General disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=48) | Control (N=48)
General Adverse Events (General disorders) | 2 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No